CLINICAL TRIAL: NCT00308607
Title: Bevacizumab, Dacarbazine and Interferon Alfa-2a Combination as a First-Line Therapy in Patients With Locally Advancing or Metastatic Melanoma
Brief Title: Bevacizumab, Dacarbazine and Interferon-Alfa to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Pia Vihinen, Turku University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 18580
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; metastatic; bevacizumab
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Bevacizumab; Dacarbazine; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab (Avastin)
Drug: dacarbazine
Drug: interferon-alfa-2a (Roferon-A)

SUMMARY:
The purpose of this study is to determine whether combination therapy with bevacizumab (Avastin), dacarbazine and interferon-alfa-2a (Roferon-A) is effective in patients with locally advancing or metastatic melanoma.

DETAILED DESCRIPTION:
Dacarbazine (DTIC) has been approved for treating metastatic melanoma in the 1970s, and after that numerous schedules and dacarbazine-based combinations have been studied in this disease. DTIC as a single agent gives a response rate of only 20%, but there have been efforts to improve this poor result by using DTIC in different combinations.Treatment of melanoma with combination chemotherapy and interferon-α (IFN-α) has given 50-60% response rates,but increase in the overall survival time has not been reached in controlled phase III studies. Thus, standard reference therapy in treatment of metastatic melanoma still is single dacarbazine or its combination with s.c. IFN-α. In addition, new studies with melanoma cells in vitro show that dacarbazine causes transcriptional up-regulation of vascular endothelial growth factor (VEGF), suggesting a potential clinical benefit of combination of DTIC and anti-VEGF therapy. IFN-α has been used in adjuvant therapy and in treatment of metastatic melanoma. IFN-α exerts its effects through antiproliferative, apoptosis-inducing and particularly antiangiogenic effects in addition to immunologic modulation.

The purpose of this study is to determine whether combination therapy with bevacizumab (Avastin), dacarbazine and interferon-alfa-2a (Roferon-A) can increase progression-free survival and overall survival in patients with locally advancing or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed malignant melanoma either locally progressing inoperable or metastatic
* measurable/evaluable disease in accordance with RECIST criteria
* WHO performance status 0-2
* normal organ function
* signed written informed consent

Exclusion Criteria:

* unevaluable disease
* major surgery within 28 days prior to day 0
* uncompleted radiotherapy
* CNS metastases
* serious non-healing wound or ulcer
* bleeding diathesis or coagulopathy
* uncontrolled hypertension
* clinically significant cardiovascular disease
* depression or psychosis, which needs medication
* ongoing treatment with aspirin (>325 mg/day)
* pregnancy
* any other serious or uncontrolled illness
* previous chemotherapy for metastatic melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Response rate according to RECIST criteria
Progression-free survival
Time to brain metastases
Overall survival

SECONDARY OUTCOMES:
To evaluate safety of this combination after every two cycles
Serum analysis of particular biochemical markers

CONTACTS AND LOCATIONS:
Overall Officials: Pia P Vihinen, MD, PhD, Principal Investigator — Turku University Hospital, Department of Oncology and Radiotherapy, Savitehtaankatu 1, FIN-20520 Turku, Finland
Locations (3):
- Finland (3):
  - Kuopio University Hospital, Kuopio, Kuopio
  - Oulu University Hospital, Oulu, Oulu
  - Tampere University Hospital, Tampere, Pirkanmaa